CLINICAL TRIAL: NCT06671847
Title: Feasibility of 24-Weeks of At-Home Chair-Based Resistance Band Training to Improve Balance, Strength, and Bone Density in Older Adults (ChaREx Study)
Brief Title: Feasibility of At-Home Chair-Based Resistance Band Training to Improve Balance, Strength, and Bone Density in Older Adults
Acronym: ChaREx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nahid Rianon, Associate Dean for Faculty Affairs, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-24-0485
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Sarcopenic Obesity
Keywords: chair-based resistance band exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Chair-based resistance band training (Experimental)
  Interventions: Device: THERABand resistance exercise bands

INTERVENTIONS:
Device: THERABand resistance exercise bands — The training will be performed using THERABand resistance exercise bands.Participants will be instructed to perform the exercises twice per week at home, for the 24 weeks duration. Each exercise session will entail 1 set of 15 repetitions of 9 different exercises

SUMMARY:
The purpose of this study is to determine the feasibility of implementing a 24-week at-home chair-based resistance band training intervention, to determine effectiveness of a the a 24-week at-home chair-based resistance band training intervention in improving body composition and to determine the effectiveness of a 24-week at-home chair-based resistance band training intervention in improving physical performance in adults 50 years and older, receiving care at the UT Physicians Center for Healthy Aging.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* receive care at the UT Physician Center for Healthy Aging

Exclusion Criteria:

* inability to provide informed consent on their own
* presence of obvious signs of cognitive decline
* a diagnosis of dementia and inability to come to the clinic for the scheduled study visits.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility as assessed by the number of people who are able to follow the prescribed exercise regimen at least 50 percent of the time | end of study (24 weeks from baseline)

SECONDARY OUTCOMES:
Change in body fat | baseline,6-months
  This will be assessed using the handheld bioelectrical impedance analysis (BIA) device (Omron HBF-510)
Change in bone mineral density (BMD) of the femoral neck and lumbar spine | baseline, 1 year from baseline
  This will be assessed by the Dual energy x-ray absorptiometry (DXA)
Handgrip strength | baseline
  This will be assessed using a validated handgrip dynamometer
Handgrip strength | 1-month
  This will be assessed using a validated handgrip dynamometer
Handgrip strength | 3-months
  This will be assessed using a validated handgrip dynamometer
Handgrip strength | 6-months
  This will be assessed using a validated handgrip dynamometer
60-second balance as assessed by the the Zibrio Stability Pro scale | Baseline
  This is determined by the patient standing on the Zibrio Stability Pro Scale unassisted for one minute and will be measured on a scale of 1 to 9 with lower scores indicating higher risk of fall
60-second balance as assessed by the the Zibrio Stability Pro scale | 1-month
  This is determined by the patient standing on the Zibrio Stability Pro Scale unassisted for one minute and will be measured on a scale of 1 to 9 with lower scores indicating higher risk of fall
60-second balance as assessed by the the Zibrio Stability Pro scale | 3-months
  This is determined by the patient standing on the Zibrio Stability Pro Scale unassisted for one minute and will be measured on a scale of 1 to 9 with lower scores indicating higher risk of fall
60-second balance as assessed by the the Zibrio Stability Pro scale | 6-months
  This is determined by the patient standing on the Zibrio Stability Pro Scale unassisted for one minute and will be measured on a scale of 1 to 9 with lower scores indicating higher risk of fall
walking gait speed | Baseline
  Gait speed will be assessed over a 6-meter distance measured within a private clinic space. The participant will be instructed to walk at their normal walking pace (as if they were walking throughout the house) and the distance/time will be converted to meters/second.Faster walking speed is related to reduced fall-risk, improved physical function, and greater survival .
walking gait speed | 1-month
  Gait speed will be assessed over a 6-meter distance measured within a private clinic space. The participant will be instructed to walk at their normal walking pace (as if they were walking throughout the house) and the distance/time will be converted to meters/second.Faster walking speed is related to reduced fall-risk, improved physical function, and greater survival .
walking gait speed | 3-months
  Gait speed will be assessed over a 6-meter distance measured within a private clinic space. The participant will be instructed to walk at their normal walking pace (as if they were walking throughout the house) and the distance/time will be converted to meters/second.Faster walking speed is related to reduced fall-risk, improved physical function, and greater survival .
walking gait speed | 6-months
  Gait speed will be assessed over a 6-meter distance measured within a private clinic space. The participant will be instructed to walk at their normal walking pace (as if they were walking throughout the house) and the distance/time will be converted to meters/second.Faster walking speed is related to reduced fall-risk, improved physical function, and greater survival .
Blood level of pro-collagen type 1 N-telopeptide (P1NP) | Baseline
  P1NP is a metabolic marker of bone formation, indicates status of bone loss and a stable or decreased level will be indicating improved metabolism
Blood level of pro-collagen type 1 N-telopeptide (P1NP) | 6 months
  P1NP is a metabolic marker of bone formation, indicates status of bone loss and a stable or decreased level will be indicating improved metabolism
Frailty as assessed by the Fried criteria | Baseline
  This consists of 5 items (unintentional weight loss, weakness [low grip strength], slowness low, self-reported exhaustion and low physical activity). Patients who meet 1or 2 of the criteria are described as pre-frail and 3 or more as frail.
Frailty as assessed by the Fried criteria | 1-month
  This consists of 5 items (unintentional weight loss, weakness [low grip strength], slowness low, self-reported exhaustion and low physical activity). Patients who meet 1or 2 of the criteria are described as pre-frail and 3 or more as frail.
Frailty as assessed by the Fried criteria | 3-months
  This consists of 5 items (unintentional weight loss, weakness [low grip strength], slowness low, self-reported exhaustion and low physical activity). Patients who meet 1or 2 of the criteria are described as pre-frail and 3 or more as frail.
Frailty as assessed by the Fried criteria | 6-months
  This consists of 5 items (unintentional weight loss, weakness [low grip strength], slowness low, self-reported exhaustion and low physical activity). Patients who meet 1or 2 of the criteria are described as pre-frail and 3 or more as frail.

CONTACTS AND LOCATIONS:
Overall Officials: Nahid Rianon, MBBS, DrPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No